CLINICAL TRIAL: NCT03624946
Title: Safety and Pharmacokinetic Evaluation of Zika Virus Immune Globulin in Healthy Volunteers
Brief Title: Study in Healthy Volunteers Evaluating Safety and Pharmacokinetics of Zika Virus Immune Globulin (ZIKV-IG)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZK-001
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Zika Virus Infection; Zika Virus Disease
Keywords: Zika virus; Human immune globulin; Hyperimmune; Polyclonal antibodies
MeSH Terms: conditions — Zika Virus Infection | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zika Virus Immune Globulin (ZIKV-IG) (Experimental): Single dose of 50 mL Zika Virus Immune Globulin (ZIKV-IG) will be administered intravenously over 33 minutes.
  Interventions: Biological: Zika Virus Immune Globulin (ZIKV-IG)
- Placebo (Saline Solution) (Placebo Comparator): Single dose of 50 mL placebo will be administered intravenously over 33 minutes.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Zika Virus Immune Globulin (ZIKV-IG) — Zika Virus Immune Globulin (ZIKV-IG) is a human immune globulin preparation containing neutralizing antibodies to Zika virus.
  Other Names: Anti-Zika Immune Globulin (Human); NP-024
  Arms: Zika Virus Immune Globulin (ZIKV-IG)
Other: Placebo — Placebo is a normal saline solution (0.9% sodium chloride).
  Other Names: Saline solution
  Arms: Placebo (Saline Solution)

SUMMARY:
Currently, there are no licensed therapeutics against Zika virus infection. Due to this unmet medical need, Zika Virus Immune Globulin (ZIKV-IG) is being developed as a therapeutic intervention against Zika virus infection. In this first-in-human study, evaluation of ZIKV-IG safety and pharmacokinetics (absorption, metabolism and excretion) will be conducted in healthy adult volunteers.

DETAILED DESCRIPTION:
This study will be evaluating safety and pharmacokinetics (PK) of one dose level of ZIKV-IG (50 mL) in healthy adult volunteers. The study is a single-center, double-blind, randomized and placebo-controlled design. The primary objective is to assess safety of intravenously (IV) administered ZIKV-IG, while the secondary objective is to determine the PK profile of ZIKV-IG in healthy adult volunteers.

There will be a total of 30 subjects enrolled into the study; dosing of the first six subjects will be staggered over three separate days, wherein two subjects per day will be randomized 1:1 to either receive 50 mL of placebo IV or 50 mL of ZIKV-IG IV (the total amount of gamma immune globulin [IgG] protein from a single 50mL dose is 4.65g). After the first six subjects are dosed, the remaining 24 subjects will be randomized 2:1 to receive either ZIKV-IG or placebo. A safety monitoring committee will review safety data (collected up to 3 days post-dosing) of the first 12 dosed subjects prior to dosing of the remaining 18 subjects. Overall, there will be 19 subjects randomized to receive ZIKV-IG and 11 subjects randomized to receive placebo on Day 1. On Day 1 (post-dose at 1 hour, 3 hours, 8 hours) and Day 2, safety and PK assessments will be conducted while the subjects are in the Phase 1 clinic. After the discharge on Day 2, the subjects will come back to the clinic for safety and PK assessments on Days 3, 4, 6, 8, 10, 12, 15, 22, 29, 43, 57 and 85. Total study duration for each subject will be up to 4 months (from screening to Day 85).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent voluntarily signed by subject.
2. Age: 18-55 years of age.
3. Blood type O+ or O-.
4. Body mass index (BMI) of 18-30.

   * Note: minimum body weight of 50 kg.
5. For female subjects (with male partners) that are not surgically sterilized (e.g., did not undergo hysterectomy, bilateral oophorectomy or tubal ligation), use of an effective method of contraception throughout the trial including:

   * Using hormonal contraception (oral, injectable or implant) continuously for 3 months prior to screening and willing to continue to use hormonal contraception throughout the entire trial.
   * Intrauterine device (IUD) inserted at least 1 month prior to screening.
   * Double barrier type of birth control measure (e.g., condoms, diaphragms, cervical sponge with spermicide).
   * True abstinence.
   * For female subjects who are post-menopausal, documented follicle- stimulating hormone (FSH) ≥40 milli-international units per milliliter (mIU/mL) must be obtained. If the FSH is <40 mIU/mL, the subject must agree to use an acceptable form of contraception (see above).
   * Females of childbearing potential without male sexual partners must be willing to maintain their sexual status as it is throughout the study.
6. For male subjects that have not had a vasectomy, use of a condom with spermicide or true abstinence for the duration of the study. Note: female partners (that are of childbearing potential) of male study subjects (that have not had a vasectomy) should use one of the effective contraception methods (eg, hormonal contraception, IUD or barrier type). Also, male subjects must not donate sperm for the duration of the study.

   * Males without female sexual partners must be willing to maintain their sexual status as it is throughout the study.
7. Healthy as determined by principal investigator or a qualified designate based on medical history, physical exam, vital signs, urinalysis, blood chemistry and hematology test results at screening.

Exclusion Criteria:

1. Use of any investigational product within the past 30 days.
2. Use of any investigational product during the study.
3. Individuals with blood type A, B or AB.
4. Recipient of any blood product within the past 12 months.
5. Plasma donation within 7 days or significant blood loss or blood donation within 56 days of baseline.
6. Blood donation at any time during the study.
7. Females with a hemoglobin level ≤120 g/L.
8. Males with a hemoglobin level <130 g/L.
9. History of hypersensitivity to blood or plasma products.
10. History of allergy to latex or rubber.
11. History of immunoglobulin A (IgA) deficiency.
12. History of hypercoagulable conditions (e.g., deep vein thrombosis or pulmonary embolism).
13. History of myocardial infarction.
14. History of stroke.
15. History of renal impairment/failure.
16. Currently pregnant or lactating or planning to become pregnant during the study.
17. History of flavivirus infection [ZIKV, dengue virus (DENV), West Nile virus (WNV), Japanese encephalitis virus (JEV), yellow fever virus (YFV)] or vaccination with licensed or investigational flavivirus vaccine.
18. Plans to travel to an area with active flavivirus (e.g., ZIKV and/or DENV) transmission during the study (and up to 10 months after the study drug administration) or has returned from an endemic area with these diseases within 30 days of screening.
19. Positive nucleic acid test (NAT) or serology for ZIKV or positive serology for WNV or DENV.
20. Positive serology test (at screening) for human immunodeficiency virus 1 and 2 (HIV), hepatitis C virus (HCV); positive test for hepatitis B virus (HBV) as determined by HBsAg.
21. History of chronic or acute severe neurologic condition (e.g., diagnosis of Guillain-Barre syndrome, epilepsy, Bell's palsy, meningitis or disease with any focal neurologic deficits).
22. Heavy smokers (≥15cigarettes a day) or electronic cigarette use.
23. History of, or suspected substance abuse problem (including alcohol).
24. Failure of drug (urine) test at screening or baseline.
25. Failure of alcohol (breath) test at screening or baseline.
26. Receipt of a live vaccine within 28 days prior to screening or anticipated receipt of a live vaccine during the study period.
27. Individuals with planned surgical procedures that will occur during the study.
28. An opinion of the investigator that it would be unwise to allow participation of the subject in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vadim Dreyzin, MD, Principal Investigator — Syneos Health; Michael McDonnell, MD, Principal Investigator — Syneos Health
Locations (1):
- Syneos Health, Early Phase, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] White J, Tunga P, Anderson DM, Iledan K, Loreth T, Parrera GS, Astacio H, Drobic B, Richardson JS. Results of a Double-Blind, Randomized, Placebo-Controlled Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Anti-Zika Virus Immunoglobulin. Am J Trop Med Hyg. 2021 Oct 4;105(6):1552-1562. doi: 10.4269/ajtmh.20-1578. PMID 34610572

RESULTS

PARTICIPANT FLOW:
Groups:
- Zika Virus Immune Globulin (ZIKV-IG): Single dose of 50 mL Zika Virus Immune Globulin (ZIKV-IG).
  Zika Virus Immune Globulin (ZIKV-IG): Zika Virus Immune Globulin (ZIKV-IG) is a human immune globulin preparation containing neutralizing antibodies to Zika virus.
Period: Overall Study
Arm/Group | Zika Virus Immune Globulin (ZIKV-IG) | Placebo (Saline Solution)
Started | 19 | 11
Completed | 19 | 10
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zika Virus Immune Globulin (ZIKV-IG) | Placebo (Saline Solution) | Total
Number analyzed (Participants) | 19 | 11 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 11 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 35 [21 to 52] | 30 [23 to 55] | 33.5 [21 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 15 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 18 | 8 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 8 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 19 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events.
Description: Number of subjects with of adverse events by severity.
Time Frame: Up to Day 85
Population: Safety population includes all subjects who received any amount of study treatment (ZIKV-IG or placebo).
Measure: Number; unit: participants
Arm/Group | Zika Virus Immune Globulin (ZIKV-IG) | Placebo (Saline Solution)
Number analyzed (Participants) | 19 | 11
participants
  Subjects with an adverse event | 12 | 8
  Subjects with a severe adverse event | 0 | 0
  Subjects with an adverse event assessed as related | 8 | 3
  Subjects with a serious adverse event | 0 | 0

2. Secondary Outcome: Assessment of Zika Virus Immune Globulin (ZIKV-IG) Maximum Concentration (Cmax)
Description: Maximum observed serum concentration of Zika Virus Immune Globulin (ZIKV-IG)
Time Frame: 0-2 hours predose to Day 85 postdose
Population: PK population included all subjects who received ZIKV-IG with adequate number of PK samples (a suitable pre-dose sample and at least one measurable post-dose sample) and PK population with subject 01-127 removed to permit comparison of the concentrations with and without the outlying subject.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/mL
Groups:
- PK Population ZIKV-IG: Subjects who received ZIKV-IG with adequate number of PK samples (a suitable pre-dose sample and at least one measurable post-dose sample), are ZIKV-negative by nucleic acid testing and serology testing and have anti-ZIKV E-protein binding antibodies <12 U/mL.
- PK Population Excluding Subject 01-127 ZIKV-IG: Subjects who received ZIKV-IG with adequate number of PK samples (a suitable pre-dose sample and at least one measurable post-dose sample), are ZIKV-negative by nucleic acid testing and serology testing and have anti-ZIKV E-protein binding antibodies <12 U/mL excluding subject 01-127.
Arm/Group | PK Population ZIKV-IG | PK Population Excluding Subject 01-127 ZIKV-IG
Number analyzed (Participants) | 19 | 18
U/mL | 171.8 (33.9) | 182.3 (21.3)

3. Secondary Outcome: Assessment of Zika Virus Immune Globulin (ZIKV-IG) Time to Maximum Concentration (Tmax)
Description: Time at which maximum serum concentration of Zika Virus Immune Globulin (ZIKV-IG) occurs.
Time Frame: 0-2 hours predose up to Day 85 postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PK Population ZIKV-IG | PK Population Excluding Subject 01-127 ZIKV-IG
Number analyzed (Participants) | 19 | 18
hours | 6.1 (16.4) | 2.3 (1.0)

4. Secondary Outcome: Assessment of Zika Virus Immune Globulin (ZIKV-IG) Area Under the Curve Up to Last Quantifiable Concentration (AUC0-t)
Description: Area under the concentration-time curve from time 0 to the last quantifiable serum Zika Virus Immune Globulin (ZIKV-IG) concentration.
Time Frame: 0-2 hours predose to Day 85 postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*U/mL
Groups:
- PK Population ZIKV-IG: Subjects who received ZIKV-IG with adequate number of PK samples (a suitable pre-dose sample and at least one measurable post-dose sample)
- PK Population Excluding Subject 01-127 ZIKV-IG: Subjects who received ZIKV-IG with adequate number of PK samples (a suitable pre-dose sample and at least one measurable post-dose sample) excluding subject 01-127 who likely did not receive the dose intravenously.
Arm/Group | PK Population ZIKV-IG | PK Population Excluding Subject 01-127 ZIKV-IG
Number analyzed (Participants) | 19 | 18
h*U/mL | 66304 (19.2) | 67221 (18.8)

5. Secondary Outcome: Assessment of Zika Virus Immune Globulin (ZIKV-IG) Area Under the Curve Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve from time 0 to the last quantifiable serum Zika Virus Immune Globulin (ZIKV-IG) concentration, plus the area extrapolated to infinity.
Time Frame: 0-2 hours predose up to Day 85 postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*U/mL
Arm/Group | PK Population ZIKV-IG | PK Population Excluding Subject 01-127 ZIKV-IG
Number analyzed (Participants) | 19 | 18
h*U/mL | 76170 (18.4) | 77224 (17.9)

6. Secondary Outcome: Assessment of Zika Virus Immune Globulin (ZIKV-IG) Clearance (CL)
Description: Total body clearance of Zika Virus Immune Globulin (ZIKV-IG) following IV administration.
Time Frame: 0-2 hours predose up to Day 85 postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | PK Population ZIKV-IG | PK Population Excluding Subject 01-127 ZIKV-IG
Number analyzed (Participants) | 19 | 18
mL/h | 6.966 (18.4) | 6.871 (17.9)

7. Secondary Outcome: Assessment of Zika Virus Immune Globulin (ZIKV-IG) Half-Life (t1/2)
Description: Apparent first order terminal elimination half-life of Zika Virus Immune Globulin (ZIKV-IG).
Time Frame: 0-2 hours predose up to Day 85 postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | PK Population ZIKV-IG | PK Population Excluding Subject 01-127 ZIKV-IG
Number analyzed (Participants) | 19 | 18
hours | 674.3 (15.9) | 674.7 (16.4)

8. Secondary Outcome: Assessment of Zika Virus Immune Globulin (ZIKV-IG) Volume of Distribution (Vz)
Description: Volume of distribution of Zika Virus Immune Globulin (ZIKV-IG) following IV administration.
Time Frame: 0-2 hours predose up to Day 85 postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | PK Population ZIKV-IG | PK Population Excluding Subject 01-127 ZIKV-IG
Number analyzed (Participants) | 19 | 18
mL | 6776.8 (20.4) | 6687.7 (20.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 (Dosing Day) through Day 85 or early withdrawal.
Description: Adverse events were unsolicited.
Arm/Group | Zika Virus Immune Globulin (ZIKV-IG) | Placebo (Saline Solution)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/11
Other Adverse Events (participants affected / at risk) | 12/19 | 8/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zika Virus Immune Globulin (ZIKV-IG) (N=19) | Placebo (Saline Solution) (N=11)
Headache (Nervous system disorders) | 4 (4) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue pigmentation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Catheter site hypoaesthesia (General disorders) | 1 (1) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Myoglobin blood increased (Investigations) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypervigilance (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the limited number of plasma donors used to generate the plasma pool for manufacture of the ZIKV-IG clinical lot, donor plasma with high isoagglutinin titers (e.g., anti-A antibodies) were not excluded from plasma pools used for the manufacture of ZIKV-IG. Therefore, in this study ZIKV-IG was for use by individuals with blood type O only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CRO agrees that Emergent shall have the exclusive right to publish the results of each Study under a Task Order, including all Work Product relating thereto, and that such results may not be published or otherwise disseminated by CRO.

DOCUMENTS (2):
  • Study Protocol (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT03624946/Prot_005.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT03624946/SAP_004.pdf